CLINICAL TRIAL: NCT05005884
Title: Evaluation of the Possible Effects of Supplement Therapy With Oral Phenolics on Plasma CD-163 Biomarker in Patients With Different Subtypes of Age-related Macular Degeneration; a Double-blind Placebo Controlled Prospective Clinical Study
Brief Title: Possible Effects of Supplement Therapy With Oral Phenolics on Cluster of Differentiation 163 (CD-163) Biomarker of Patients With Age-related Macular Degeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Swiss Eye Institute (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1401
Record Dates: First submitted 2021-08-01; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral phenolics intake (Active Comparator): Prescription of oral phenolics 250 mg two times daily
  Interventions: Drug: Oral intake of medication
- placebo caplet intake (Placebo Comparator): Prescription of oral phenolics 250 mg two times daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral intake of medication — Prescription of oral phenolics 250 mg two times daily
  Arms: oral phenolics intake
Drug: Placebo — Prescription of oral phenolics 250 mg two times daily
  Arms: placebo caplet intake

SUMMARY:
In this multi-center study, possible effects of supplement treatment with oral phenolics on plasma CD-163 and progression of dry and wet age-related macular degeneration (AMD) via evaluating the CD163 before and after the prescription of this drug will be evaluated in patients with dry type AMD and Neo vascular age-related macular degeneration (nAMD).

Both AMD subgroups will be recruited. In terms of evaluation of the effects of phenolics (500 mg caplets/day) on AMD progression, patients will be randomized and divided into 2 subgroups i.e. (i) receiving phenolics supplementation; and, (ii) receiving placebo for 1 month. The phenolics/placebo caplets will resemble completely and be encoded at origin; Neither the participants nor the researchers will be informed about the codes until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of intermediate to late AMD (dry AMD and nAMD )
* Age-matched controls without any sign of AMD
* Signed informed consent

Exclusion Criteria:

* Systemic disease or other eye-related diseases (diabetes, immunologic or inflammatory, active or chronic infectious disease, active malignancy, uveitis, retinal vascular occlusive disease, glaucoma)
* Systemic therapy with corticosteroids or biological drugs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Plasma CD-163 | 1 month
  Blood sampling

SECONDARY OUTCOMES:
Decimal acuity of vision | 1 month
  Snellen chart

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran